CLINICAL TRIAL: NCT01443013
Title: Predictive Value Analysis of Messenger Ribonucleic Acid (mRNA) Urinary Expression of Foxp3 and Vimentin on Graft Outcome in Renal Transplant Recipient: National Prospective Study
Brief Title: Analysis of Foxp3 and Vimentin Expression in Renal Transplant Recipient
Acronym: TUFEV
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI08031; AOM09031 (Other: Other sponsor number)
Record Dates: First submitted 2011-08-09; First posted 2011-09-29 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Function of Renal Transplant
Keywords: Tolerance; Renal Transplantation; Chronic allograft nephropathy
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine for mRNA extraction and congelation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cohort of Renal Transplant recipients
  Interventions: Other: Renal Transplant

INTERVENTIONS:
Other: Renal Transplant — urinary sample at month 3, 6 and 12

SUMMARY:
This observational study is designed to analyse the urinary mRNA expression of Foxp3 and Vimentin, two genes involved in tolerance and early graft dysfunction in 500 renal transplant recipients from 17 renal transplant site in France and to determine the predictive value of these gene expression on the one year graft outcome including graft function, one-year graft histological analysis and incidence of acute rejection.

DETAILED DESCRIPTION:
This observational study is designed to analyse the urinary mRNA expression of Foxp3 and Vimentin, two genes involved in tolerance and early graft dysfunction in 500 renal transplant recipients from 17 renal transplant site in France and to determine the predictive value of these gene expression on the one year graft outcome including graft function,

ELIGIBILITY:
Inclusion Criteria:

* All renal transplant recipients aged >18 years with informed consent
* Kidney transplantation in one of the centers participating in the study all patients registered on the waiting list to the Agency of Biomedicine
* Supported by a conventional procedure
* Informed consent signed.
* No pregnancy or lactation in progress.
* Serology HIV and (HCV negative suppressed by amendment n°2)
* No contraindication for a biopsy at 1 year post transplant

Exclusion Criteria:

* Positive crossmatch, focal segmental glomerulosclerosis (FSGS) as primary nephropathy, HIV positive population
* Absence of registration on the waiting list for transplantation with the Agency of Biomedicine
* HIV-positive serology
* Chronic renal failure secondary to focal segmental hyalinosis
* Cross-match historical or cross match of the day positive T or B awareness
* Patient included in a Memorandum of industry (suppressed by amendment n°1)
* No affiliation to a social security scheme
* Patients with early failure due to immediate complications (4%) will be included but will not be considered for analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Foxp3 and Vimentin mRNA expression | at Month 1,3,6 and 12
  evaluation at month 9 suppressed by amendment n°2

SECONDARY OUTCOMES:
Renal biopsy | at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Grimbert, MD PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Aquino-Dias EC, Joelsons G, da Silva DM, Berdichevski RH, Ribeiro AR, Veronese FJ, Goncalves LF, Manfro RC. Non-invasive diagnosis of acute rejection in kidney transplants with delayed graft function. Kidney Int. 2008 Apr;73(7):877-84. doi: 10.1038/sj.ki.5002795. Epub 2008 Jan 23. PMID 18216781